CLINICAL TRIAL: NCT03054337
Title: Phase 2, Randomized, Double-Blind, Placebo Controlled, Dose-Finding Study to Assess the Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics of Vadadustat in Japanese Subjects With Anemia Secondary to Non-Dialysis Dependent Chronic Kidney Disease (NDD-CKD)
Brief Title: Dose-Finding Study of Vadadustat in Japanese Subjects With Anemia Secondary to Non-Dialysis Dependent Chronic Kidney Disease (NDD-CKD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0021
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Anemia; Non-dialysis Dependent Chronic Kidney Disease
Keywords: Anemia; kidney; non-dialysis dependent chronic kidney disease; CKD; NDD-CKD; renal; vadadustat; AKB-6548; hypoxia-inducible factor; hypoxia-inducible factor (HIF); HIF; prolyl-hydroxylase inhibitor (PHI); PHI; Japan; Japanese; Akebia (AKB)
MeSH Terms: conditions — Anemia | interventions — vadadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Vadadustat, Dose 1 (Experimental): Daily oral dose
  Interventions: Drug: Vadadustat
- Vadadustat, Dose 2 (Experimental): Daily oral dose
  Interventions: Drug: Vadadustat
- Vadadustat, Dose 3 (Experimental): Daily oral dose
  Interventions: Drug: Vadadustat
- Placebo (Placebo Comparator): Daily oral dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vadadustat
  Other Names: AKB-6548
  Arms: Vadadustat, Dose 1; Vadadustat, Dose 2; Vadadustat, Dose 3
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, dose-finding study to assess the efficacy, safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) of orally administered vadadustat in Japanese participants with anemia secondary to Non-dialysis Dependent Chronic Kidney Disease (NDD-CKD).

ELIGIBILITY:
Inclusion Criteria:

* Male and female Japanese participants ≥20 years of age
* Diagnosis of chronic kidney disease (CKD) based on an estimated glomerular filtration rate ≤60 milliliters per minute per 1.73 meters squared (mL/min/1.73 m^2)
* Hemoglobin (Hb) ≤10.5 grams per deciliter (g/dL)
* Not currently being treated with dialysis and not expected to start dialysis within 3 months of screening

Exclusion Criteria:

* Anemia due to a cause other than CKD or presence of active bleeding or recent blood loss
* Sickle cell disease, myelodysplastic syndromes, bone marrow fibrosis, hematologic malignancy, myeloma, hemolytic anemia, thalassemia, or pure red cell aplasia
* Red blood cell transfusion within 4 weeks prior to or during screening
* Intravenous iron within 4 weeks prior to or during screening
* Any use of erythropoiesis-stimulating agents within 6 weeks prior to or during screening

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Sponsor GmbH
Locations (18):
- Japan (18):
  - Aichi
  - Chiba
  - Ehime
  - Gunma
  - Hiroshima
  - Hokkaido
  - Hyōgo
  - Ibaraki
  - Kanagawa
  - Nagano
  - Nara
  - Niigata
  - Okayama
  - Okinawa
  - Osaka
  - Ōita
  - Shiga
  - Tokushima

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Groups:
- Vadadustat 150 mg: Participants were randomized to receive vadadustat 150 milligrams (mg), administered as 1 tablet once daily (QD), for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target hemoglobin (Hb) of 10.0 to 12.0 grams/deciliter (g/dL) based on dose adjustment guidelines.
- Vadadustat 300 mg: Participants were randomized to receive vadadustat 300 mg, administered as 2 tablets QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Vadadustat 600 mg: Participants were randomized to receive vadadustat 600 mg, administered as 4 tablets QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Placebo to Vadadustat 150 mg: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 150 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Placebo to Vadadustat 300 mg: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 300 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Placebo to Vadadustat 600 mg: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 600 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
Period: Primary Efficacy Period (6 Weeks)
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Started | 12 | 12 | 13 | 5 | 4 | 5
Completed | 12 | 12 | 13 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Adjustment and Maintenance Period
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Started | 12 | 12 | 13 | 5 | 4 | 5
Completed | 11 | 10 | 12 | 5 | 4 | 4
Not Completed | 1 | 2 | 1 | 0 | 0 | 1
Not completed — Investigator discretion | 1 | 2 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Safety Population, comprised of all enrolled participants who received at least 1 dose of study medication. The Safety Population was based on the actual treatment that participants received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg | Total
Number analyzed (Participants) | 12 | 12 | 13 | 5 | 4 | 5 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (10.33) | 65.8 (11.53) | 71.5 (12.84) | 73.4 (3.05) | 68.0 (21.21) | 72.2 (8.64) | 70.2 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 8 | 1 | 1 | 2 | 22
  Male | 7 | 7 | 5 | 4 | 3 | 3 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hemoglobin Levels [Mean (Standard Deviation); unit: grams per deciliter (g/dL)] | 9.958 (0.8051) | 9.492 (0.8867) | 9.500 (0.8446) | 10.280 (0.9365) | 9.625 (0.6551) | 9.680 (0.8198) | 9.710 (0.8410)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin (Hb) Levels From Pre-treatment to the End of the Primary Efficacy Period
Description: The pre-treatment value for Hb was defined as the average of 2 values obtained prior to treatment, i.e., the qualifying screening value and the Baseline value. Change from Pre-treatment was calculated as the Week 6 value minus the Pre-treatment value.
Time Frame: Pre-treatment; Week 6
Population: Modified Intent-to-Treat Population (mITT): all randomized participants who received at least 1 dose of study medication, had a pre-treatment Hb average, and at least one post-Baseline Hb measurement. The mITT Population was based on the treatment to which participants were randomized.
Measure: Least Squares Mean (Standard Error); unit: grams per deciliter (g/dL)
Groups:
- Vadadustat 150: Participants were randomized to receive vadadustat 150 milligrams (mg), administered as 1 tablet once daily (QD), for 6 weeks.
- Vadadustat 300 mg: Participants were randomized to receive vadadustat 300 mg, administered as 2 tablets QD, for 6 weeks.
- Vadadustat 600 mg: Participants were randomized to receive vadadustat 600 mg, administered as 4 tablets QD, for 6 weeks.
- Placebo: Participants were randomized to receive matching placebo for 6 weeks.
Arm/Group | Vadadustat 150 | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 14
grams per deciliter (g/dL) | 0.43 (0.224) | 1.13 (0.223) | 1.62 (0.215) | -0.47 (0.206)
Statistical Analysis 1: Comparison: Vadadustat 150 vs Placebo; Test type: Superiority; p = 0.0045, ANCOVA; The analysis of covariance (ANCOVA) model included treatment assignment (3 dosed groups; 1 placebo group) and pre-treatment Hb value as a covariate; Least squares mean difference = 0.90, 95% CI 2-sided [0.29 to 1.51], Standard Error of Mean 0.301
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment assignment (3 dosed groups; 1 placebo group) and pre-treatment Hb value as a covariate; Least squares mean difference = 1.59, 95% CI 2-sided [0.98 to 2.21], Standard Error of Mean 0.306
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 2]; Least squares mean difference = 2.09, 95% CI 2-sided [1.49 to 2.70], Standard Error of Mean 0.300

2. Secondary Outcome: Time to Reach the Target Hb Level of 10.0 to 12.0 g/dL From Baseline up to Week 16
Description: Time for this analysis was measured from Day 1 (Baseline) through the point in time during either the Primary Efficacy Period or the Dose Adjustment and Maintenance Period when a participant's Hb level achieved the target range of 10.0 to 12.0 g/dL.
Time Frame: from Baseline up to Week 16
Population: mITT Population. Only participants with Hb < 10.0 g/dL at the Baseline visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Vadadustat 150 mg: Participants were randomized to receive vadadustat 150 mg, administered as 1 tablet QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target hemoglobin (Hb) of 10.0 to 12.0 grams/deciliter (g/dL) based on dose adjustment guidelines.
- Vadadustat 600 mg: Participants were randomized to receive vadadustat 600 mg, administered as 4 tablets OD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target hemoglobin of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 6 | 7 | 8 | 2 | 3 | 4
days | 56.8 (43.31) | 39.0 (38.52) | 25.6 (16.47) | 79.0 (11.31) | 71.0 (14.00) | 54.5 (33.67)

3. Secondary Outcome: Mean Hb Levels at the End of the Primary Efficacy Period
Description: Data are reported as mean of the actual Week 6 values.
Time Frame: up to Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Vadadustat 150 mg: Participants were randomized to receive vadadustat 150 mg, administered as 1 tablet QD, for 6 weeks.
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 14
g/dL | 10.392 (0.7280) | 10.675 (1.2693) | 11.162 (1.1169) | 9.421 (0.9242)

4. Secondary Outcome: Mean Hb Levels at the End of the Dose Adjustment and Maintenance Period
Description: Data are reported as mean of the actual Week 16 values.
Time Frame: up to Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Vadadustat 150 mg: Participants were randomized to receive vadadustat 150 mg, administered as 1 tablet QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 11 | 10 | 12 | 5 | 4 | 4
g/dL | 10.973 (0.5711) | 11.230 (0.7514) | 11.342 (0.6473) | 10.860 (0.5857) | 11.425 (0.9179) | 11.950 (0.6608)

5. Secondary Outcome: Number of Participants Who Achieved the Target Hb Level of 10.0 to 12.0 g/dL at the End of the Dose Adjustment and Maintenance Period
Time Frame: up to Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 11 | 10 | 12 | 5 | 4 | 4
Participants | 11 | 8 | 11 | 5 | 3 | 2

6. Secondary Outcome: Mean Change in Hb Between Pre-treatment and the End of the Dose Adjustment and Maintenance Period
Description: The pre-treatment value for Hb was defined as the average of 2 values obtained prior to treatment, i.e., the qualifying screening value and the Baseline value. Change from Pre-treatment was calculated as the Week 16 value minus the Pre-treatment value.
Time Frame: Pre-treatment; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 11 | 10 | 12 | 5 | 4 | 4
g/dL | 0.982 (0.3676) | 1.610 (1.1692) | 1.779 (0.8117) | 0.790 (0.3070) | 1.538 (0.5250) | 2.075 (0.2784)

7. Secondary Outcome: Mean Change in Red Blood Cell (RBC) Count and Absolute Reticulocyte Count From Baseline to the End of the Primary Efficacy Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: 10^6 cells/microliter (μL)
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 14
10^6 cells/microliter (μL)
  RBC Count | 0.17 (0.075) | 0.34 (0.075) | 0.48 (0.073) | -0.17 (0.070)
  Absolute Reticulocyte Count | 0.01 (0.004) | 0.01 (0.003) | 0.01 (0.003) | 0.01 (0.003)
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; RBC Count; Test type: Superiority; p = 0.0018, ANCOVA; The ANCOVA model will include treatment assignment (3 dosed groups; 1 placebo group) and pre-treatment Hb value as a covariate; Least squares mean difference = 0.34, 95% CI 2-sided [0.13 to 0.55], Standard Error of Mean 0.103
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; RBC Count; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = 0.51, 95% CI 2-sided [0.30 to 0.72], Standard Error of Mean 0.103
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; RBC Count; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = 0.66, 95% CI 2-sided [0.45 to 0.86], Standard Error of Mean 0.102
Statistical Analysis 4: Comparison: Vadadustat 150 mg vs Placebo; Absolute Reticulocyte Count; Test type: Superiority; p = 0.7804, ANCOVA; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = 0.00, 95% CI 2-sided [-0.01 to 0.01], Standard Error of Mean 0.005
Statistical Analysis 5: Comparison: Vadadustat 300 mg vs Placebo; Absolute Reticulocyte Count; Test type: Superiority; p = 0.0986, ANCOVA; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = 0.01, 95% CI 2-sided [-0.00 to 0.02], Standard Error of Mean 0.005
Statistical Analysis 6: Comparison: Vadadustat 600 mg vs Placebo; Absolute Reticulocyte Count; Test type: Superiority; p = 0.1661, ANCOVA; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = 0.01, 95% CI 2-sided [-0.00 to 0.02], Standard Error of Mean 0.005

8. Secondary Outcome: Mean Change in RBC Count and Absolute Reticulocyte Count From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^6 cells/μL
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 11 | 10 | 12 | 5 | 4 | 4
10^6 cells/μL
  RBC Count | 0.305 (0.1870) | 0.476 (0.4406) | 0.593 (0.3186) | 0.186 (0.2165) | 0.438 (0.2175) | 0.608 (0.1771)
  Absolute Reticulocyte Count | 0.003078 (0.0094008) | 0.008001 (0.0156884) | 0.000196 (0.0085029) | 0.010716 (0.0279909) | 0.009703 (0.0103348) | 0.000595 (0.0171563)

9. Secondary Outcome: Mean Change in Hematocrit and Reticulocytes From Baseline to the End of the Primary Efficacy Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 14
percentage
  Hematocrit | 2.13 (0.696) | 4.13 (0.696) | 6.07 (0.667) | -1.17 (0.643)
  Reticulocytes | 0.16 (0.111) | 0.28 (0.111) | 0.19 (0.107) | 0.25 (0.103)
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; Hematocrit; Test type: Superiority; p = 0.0010, ANCOVA; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = 3.30, 95% CI 2-sided [1.40 to 5.20], Standard Error of Mean 0.942
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; Hematocrit; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = 5.30, 95% CI 2-sided [3.38 to 7.22], Standard Error of Mean 0.953
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; Hematocrit; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = 7.24, 95% CI 2-sided [5.37 to 9.11], Standard Error of Mean 0.930
Statistical Analysis 4: Comparison: Vadadustat 150 mg vs Placebo; Reticulocytes; Test type: Superiority; p = 0.5889, ANCOVA; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = -0.08, 95% CI 2-sided [-0.39 to 0.22], Standard Error of Mean 0.152
Statistical Analysis 5: Comparison: Vadadustat 300 mg vs Placebo; Reticulocytes; Test type: Superiority; p = 0.8074, ANCOVA; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = 0.04, 95% CI 2-sided [-0.27 to 0.34], Standard Error of Mean 0.151
Statistical Analysis 6: Comparison: Vadadustat 600 mg vs Placebo; Reticulocytes; Test type: Superiority; p = 0.6952, ANCOVA; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = -0.06, 95% CI 2-sided [-0.36 to 0.24], Standard Error of Mean 0.148

10. Secondary Outcome: Mean Change in Hematocrit and Reticulocytes From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 11 | 10 | 12 | 5 | 4 | 4
percentage
  Hematocrit | 3.28 (1.947) | 5.17 (4.991) | 5.39 (2.844) | 2.32 (1.827) | 5.80 (1.566) | 6.05 (1.997)
  Reticulocytes | -0.02 (0.232) | 0.07 (0.442) | -0.18 (0.279) | 0.28 (0.893) | 0.15 (0.238) | -0.18 (0.377)

11. Secondary Outcome: Mean Change in Iron and Total Iron Binding Capacity (TIBC) From Baseline to the End of the Primary Efficacy Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: mITT Population
Measure: Mean (Standard Deviation); unit: micrograms per deciliter (μg/dL)
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 14
micrograms per deciliter (μg/dL)
  Iron | -1.8 (19.58) | -2.4 (20.75) | 4.4 (30.82) | -7.4 (19.92)
  TIBC | 44.9 (32.9) | 75.2 (35.60) | 93.8 (44.74) | 7.6 (23.55)
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; Iron; Test type: Superiority; p = 0.3702, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; Iron; Test type: Superiority; p = 0.5524, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; Iron; Test type: Superiority; p = 0.1589, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 4: Comparison: Vadadustat 150 mg vs Placebo; TIBC; Test type: Superiority; p = 0.0092, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 5: Comparison: Vadadustat 300 mg vs Placebo; TIBC; Test type: Superiority; p < 0.0001, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 6: Comparison: Vadadustat 600 mg vs Placebo; TIBC; Test type: Superiority; p < 0.0001, ANCOVA; test of treatment group difference based on ANCOVA model

12. Secondary Outcome: Mean Change in Iron and TIBC From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 11 | 10 | 12 | 5 | 4 | 4
μg/dL
  Iron | 11.7 (38.25) | 3.5 (31.17) | 11.5 (28.56) | -1.4 (21.82) | 5.5 (24.66) | 5.8 (25.59)
  TIBC | 51.8 (48.41) | 43.4 (42.77) | 42.8 (28.28) | 47.6 (21.71) | 73.5 (39.95) | 44.5 (43.19)

13. Secondary Outcome: Mean Change in Transferrin Saturation (TSAT) From Baseline to the End of the Primary Efficacy Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 14
percentage | -4.96 (7.343) | -7.31 (8.380) | -6.78 (10.609) | -4.72 (8.931)
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; Test type: Superiority; p = 0.9092, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; Test type: Superiority; p = 0.1484, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; Test type: Superiority; p = 0.1313, ANCOVA; test of treatment group difference based on ANCOVA model

14. Secondary Outcome: Mean Change in TSAT From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 11 | 10 | 12 | 5 | 4 | 4
percentage | -1.47 (10.365) | -2.68 (13.201) | -0.19 (9.857) | -7.00 (12.247) | -5.03 (11.342) | -2.68 (10.608)

15. Secondary Outcome: Mean Change in Ferritin and Hepcidin From Baseline to the End of the Primary Efficacy Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 14
nanograms per milliliter (ng/mL)
  Ferritin | -38.48 (34.227) | -69.36 (49.965) | -101.54 (57.697) | -11.44 (31.408)
  Hepcidin | -24.622 (20.0165) | -40.819 (27.2486) | -37.964 (21.0819) | -3.824 (18.4986)
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; Ferritin; Test type: Superiority; p = 0.1080, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 2: Comparison: Vadadustat 300 mg vs Placebo; Ferritin; Test type: Superiority; p = 0.0002, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 3: Comparison: Vadadustat 600 mg vs Placebo; Ferritin; Test type: Superiority; p < 0.0001, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 4: Comparison: Vadadustat 150 mg vs Placebo; Hepcidin; Test type: Superiority; p = 0.0672, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 5: Comparison: Vadadustat 300 mg vs Placebo; Hepcidin; Test type: Superiority; p = 0.0004, ANCOVA; test of treatment group difference based on ANCOVA model
Statistical Analysis 6: Comparison: Vadadustat 600 mg vs Placebo; Hepcidin; Test type: Superiority; p < 0.0001, ANCOVA; test of treatment group difference based on ANCOVA model

16. Secondary Outcome: Mean Change in Ferritin and Hepcidin From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 11 | 10 | 12 | 5 | 4 | 4
ng/mL
  Ferritin | -79.45 (39.655) | -62.35 (36.808) | -59.68 (59.843) | -69.26 (46.519) | -146.63 (34.261) | -59.43 (13.618)
  Hepcidin | -29.522 (22.7101) | -23.061 (53.0161) | -2.502 (21.2660) | -9.464 (19.1361) | -38.920 (23.4788) | -9.745 (9.2100)

17. Secondary Outcome: Number of Participants Who Required Rescue With Erythropoiesis-stimulating Agents (ESAs) From Baseline to the End of the Primary Efficacy Period
Description: ESA rescue is defined as participants with ESA administration and 1) the participant experienced a clinically significant worsening of their anemia or symptoms of anemia, 2) the participant's Hb level is <9.0 g/dL, and 3) reason for early study withdrawal of worsening of anemia requiring ESA rescue or blood transfusion. Participants who initiated rescue therapy (including ESAs) were required to stop study drug treatment and were discontinued from the study.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 14
Participants | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants Who Required Rescue With ESAs From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: as for outcome 17
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 12 | 12 | 13 | 5 | 4 | 5
Participants | 0 | 2 | 1 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants Who Required Rescue With a RBC Transfusion From Baseline to the End of the Primary Efficacy Period
Description: Participants who initiated rescue therapy (including RBC transfusion) were required to stop study drug treatment and were discontinued from the study.
Time Frame: Baseline; Week 6
Population: mITT Population. Only participant with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 14
Participants | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants Who Required Rescue With a RBC Transfusion From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: as for outcome 19
Time Frame: Baseline; Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 12 | 12 | 13 | 5 | 4 | 5
Participants | 0 | 1 | 1 | 0 | 0 | 1

21. Secondary Outcome: Number of the Participants With the Indicated Number of Dose Adjustments From Baseline to the End of the Dose Adjustment and Maintenance Period
Description: Increases in dose were not allowed during the 6-week Primary Efficacy Period.
Time Frame: Baseline to Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 12 | 12 | 13 | 5 | 4 | 5
Participants
  0 dose adjustments | 3 | 1 | 2 | 0 | 0 | 1
  1 dose adjustment | 5 | 7 | 1 | 3 | 1 | 1
  2 dose adjustments | 3 | 4 | 3 | 1 | 1 | 2
  3 or more dose adjustments | 1 | 0 | 7 | 1 | 2 | 1

22. Secondary Outcome: Number of Participants Who Maintained Iron Sufficiency From Baseline to Week 6
Description: Iron sufficiency was defined as ferritin ≥50 ng/mL and TSAT ≥20%.
Time Frame: Baseline to Week 6
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 14
Participants
  Iron sufficiency maintained | 7 | 4 | 4 | 9
  Iron sufficiency not maintained | 5 | 8 | 9 | 5
Statistical Analysis 1: Comparison: Vadadustat 150 mg vs Placebo; Test type: Superiority; p = 0.0895, Fisher Exact
Statistical Analysis 2: Comparison: Vadadustat 300 mg; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Vadadustat 600 mg; Test type: Superiority; p = 0.3845, Fisher Exact

23. Secondary Outcome: Number of Participants Who Maintained Iron Sufficiency From Baseline to Week 16
Description: Iron sufficiency was defined as ferritin ≥50 ng/mL and TSAT ≥20%.
Time Frame: Baseline to Week 16
Population: mITT Population. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 12 | 12 | 13 | 5 | 4 | 5
Participants
  Iron sufficiency maintained | 6 | 2 | 4 | 1 | 1 | 0
  Iron sufficiency not maintained | 6 | 10 | 9 | 4 | 3 | 5

24. Secondary Outcome: Plasma Concentration Profile of Vadadustat and Its Metabolites Using a Pre-dose Sample From Week 4
Description: Blood samples were collected for analysis.
Time Frame: Week 4, pre-dose
Population: Pharmacokinetic (PK) Population: all participants in the Safety Population (all enrolled participants who received at least 1 dose of study medication) who had a pre-dose PK sample at Week 4.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 0
micrograms per milliliter (µg/mL)
  Vadadustat | 5530.9 (4168.86) | 12955.8 (9771.65) | 19291.5 (9325.30) |
  O-glucuronide | 3914.7 (5772.39) | 12358.6 (7586.73) | 16586.2 (12363.44) |
  Acyl-glucuronide | 0.00 (0.000) | 1.95 (6.755) | 8.99 (16.430) |

25. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (SAEs) in the Primary Efficacy Period
Description: An adverse event (AE) was defined as any untoward medical occurrence (including a clinically significant abnormal laboratory finding) that occurred in the protocol-specified AE reporting period. An AE included medical conditions, signs, and symptoms not previously observed in the participant that emerged during the protocol-specified AE reporting period, including signs or symptoms associated with pre-existing underlying conditions that were not present prior to the AE reporting period. An AE that met one or more of the following criteria or outcomes was classified as serious: death; life-threatening; in-patient hospitalization or prolongation of existing hospitalization; persistent or significant disability/ incapacity; congenital anomaly/birth defect; was considered a medically important event not meeting the above criteria, but which could jeopardize a participant, or could require medical or surgical intervention to prevent one of the criteria listed in this definition.
Time Frame: up to Week 6
Population: Safety Population: all enrolled participants who received at least 1 dose of study medication. The Safety Population was based on the actual treatment that participants received.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 14
Participants
  TEAEs | 4 | 7 | 7 | 5
  Treatment-emergent SAEs | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Participants With TEAEs and Treatment-emergent SAEs in the Dose Adjustment and Maintenance Period
Description: An AE was defined as any untoward medical occurrence (including a clinically significant abnormal laboratory finding) that occurred in the protocol-specified AE reporting period. An AE included medical conditions, signs, and symptoms not previously observed in the participant that emerged during the protocol-specified AE reporting period, including signs or symptoms associated with pre-existing underlying conditions that were not present prior to the AE reporting period. An AE that met one or more of the following criteria or outcomes was classified as serious: death; life-threatening; in-patient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; was considered a medically important event not meeting the above criteria, but which could jeopardize a participant, or could require medical or surgical intervention to prevent one of the criteria listed in this definition.
Time Frame: up to Week 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat 150 mg | Vadadustat 300 mg | Vadadustat 600 mg | Placebo to Vadadustat 150 mg | Placebo to Vadadustat 300 mg | Placebo to Vadadustat 600 mg
Number analyzed (Participants) | 12 | 12 | 13 | 5 | 4 | 5
Participants
  TEAEs | 9 | 10 | 6 | 3 | 3 | 3
  Treatment-emergent SAEs | 0 | 5 | 2 | 1 | 1 | 2

ADVERSE EVENTS:
Time Frame: up to Week 18
Groups:
- Primary Efficacy Period: 150 mg Vadadustat: Participants were randomized to receive vadadustat 150 milligrams (mg), administered as 1 tablet once daily (QD), for 6 weeks.
- Primary Efficacy Period: 300 mg Vadadustat: Participants were randomized to receive vadadustat 300 mg, administered as 2 tablets QD, for 6 weeks.
- Primary Efficacy Period: 600 mg Vadadustat: Participants were randomized to receive vadadustat 600 mg, administered as 4 tablets QD, for 6 weeks.
- Primary Efficacy Period: Placebo Matched to 150 mg Vadadustat; Primary Efficacy Period: Placebo Matched to 300 mg Vadadustat; Primary Efficacy Period: Placebo Matched to 600 mg Vadadustat: Participants were randomized to receive matching placebo for 6 weeks.
- Dose Adjustment and Maintenance: 150 mg Vadadustat: Participants were randomized to receive vadadustat 150 mg, administered as 1 tablet QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target hemoglobin (Hb) of 10.0 to 12.0 grams per deciliter (g/dL) based on dose adjustment guidelines.
- Dose Adjustment and Maintenance: 300 mg Vadadustat: Participants were randomized to receive vadadustat 300 mg, administered as 2 tablets QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Dose Adjustment and Maintenance: 600 mg Vadadustat: Participants were randomized to receive vadadustat 600 mg, administered as 4 tablets QD, for 6 weeks during the Primary Efficacy Period. During the 10-week Dose Adjustment and Maintenance Period, the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Dose Adjustment and Maintenance: Placebo to 150 mg Vadadustat: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period.
  During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 150 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Dose Adjustment and Maintenance: Placebo to 300 mg Vadadustat: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period.
  During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 300 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
- Dose Adjustment and Maintenance: Placebo to 600 mg Vadadustat: Participants were randomized to receive matching placebo for 6 weeks during the Primary Efficacy Period.
  During the 10-week Dose Adjustment and Maintenance Period, participants randomized to receive placebo in the 6-week Efficacy Period were switched to vadadustat 600 mg, and the dose was adjusted to achieve a target Hb of 10.0 to 12.0 g/dL based on dose adjustment guidelines.
Arm/Group | Primary Efficacy Period: 150 mg Vadadustat | Primary Efficacy Period: 300 mg Vadadustat | Primary Efficacy Period: 600 mg Vadadustat | Primary Efficacy Period: Placebo Matched to 150 mg Vadadustat | Primary Efficacy Period: Placebo Matched to 300 mg Vadadustat | Primary Efficacy Period: Placebo Matched to 600 mg Vadadustat | Dose Adjustment and Maintenance: 150 mg Vadadustat | Dose Adjustment and Maintenance: 300 mg Vadadustat | Dose Adjustment and Maintenance: 600 mg Vadadustat | Dose Adjustment and Maintenance: Placebo to 150 mg Vadadustat | Dose Adjustment and Maintenance: Placebo to 300 mg Vadadustat | Dose Adjustment and Maintenance: Placebo to 600 mg Vadadustat
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/5 | 0/4 | 0/5 | 0/12 | 0/12 | 0/13 | 0/5 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/5 | 0/4 | 0/5 | 0/12 | 5/12 | 2/13 | 1/5 | 1/4 | 2/5
Other Adverse Events (participants affected / at risk) | 4/12 | 7/12 | 7/13 | 0/5 | 2/4 | 3/5 | 9/12 | 10/12 | 6/13 | 2/5 | 2/4 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Efficacy Period: 150 mg Vadadustat (N=12) | Primary Efficacy Period: 300 mg Vadadustat (N=12) | Primary Efficacy Period: 600 mg Vadadustat (N=13) | Primary Efficacy Period: Placebo Matched to 150 mg Vadadustat (N=5) | Primary Efficacy Period: Placebo Matched to 300 mg Vadadustat (N=4) | Primary Efficacy Period: Placebo Matched to 600 mg Vadadustat (N=5) | Dose Adjustment and Maintenance: 150 mg Vadadustat (N=12) | Dose Adjustment and Maintenance: 300 mg Vadadustat (N=12) | Dose Adjustment and Maintenance: 600 mg Vadadustat (N=13) | Dose Adjustment and Maintenance: Placebo to 150 mg Vadadustat (N=5) | Dose Adjustment and Maintenance: Placebo to 300 mg Vadadustat (N=4) | Dose Adjustment and Maintenance: Placebo to 600 mg Vadadustat (N=5)
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
End-stage renal disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arteriovenous shunt procedure (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Efficacy Period: 150 mg Vadadustat (N=12) | Primary Efficacy Period: 300 mg Vadadustat (N=12) | Primary Efficacy Period: 600 mg Vadadustat (N=13) | Primary Efficacy Period: Placebo Matched to 150 mg Vadadustat (N=5) | Primary Efficacy Period: Placebo Matched to 300 mg Vadadustat (N=4) | Primary Efficacy Period: Placebo Matched to 600 mg Vadadustat (N=5) | Dose Adjustment and Maintenance: 150 mg Vadadustat (N=12) | Dose Adjustment and Maintenance: 300 mg Vadadustat (N=12) | Dose Adjustment and Maintenance: 600 mg Vadadustat (N=13) | Dose Adjustment and Maintenance: Placebo to 150 mg Vadadustat (N=5) | Dose Adjustment and Maintenance: Placebo to 300 mg Vadadustat (N=4) | Dose Adjustment and Maintenance: Placebo to 600 mg Vadadustat (N=5)
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema due to renal disease (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angular cheilitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Parathyroid gland enlargement (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT03054337/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT03054337/SAP_001.pdf